CLINICAL TRIAL: NCT05691855
Title: 89Zr-labeled NY009 PET Imaging in Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Jiangnan University (Other)
Responsible Party: Principal Investigator, Chunjing Yu, Director, Affiliated Hospital of Jiangnan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2020002
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2022-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 89Zr-NY009 (Experimental)
  Interventions: Drug: 89Zr-NY009

INTERVENTIONS:
Drug: 89Zr-NY009 — Patients will receive a tracer (5-10mg, IV) dose of 89Zr (2-3mCi) labelled NY009

SUMMARY:
This is a single arm study to evaluate the safety and biodistribution of 89Zr-labeled NY009 PET Imaging in patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily signed informed consent;
2. Age 18-75, male or female;
3. Patients diagnosed with cancer confirmed by histopathology or cytology;
4. At least one measurable solid lesion has been examined according RECIST1.1 standard;
5. ECOG score 0~2.

Exclusion Criteria:

1. Recovery from major trauma (including surgery) within 4 weeks prior to study treatment;
2. Patients with systemic or locally severe infections, or other serious coexisting diseases;
3. Patients with abnormal immune function or who have recently used immunosuppressive or potentiating agents including various vaccines;
4. Patients with autoimmune diseases, including rheumatoid arthritis;
5. Inadequate control of arrhythmias, including atrial fibrillation;
6. Uncontrolled hypertension;
7. Patients with allergies or allergies to any component of the imaging agent or antibody;
8. Patients who cannot undergo PET/CT imaging scan;
9. Syphilis, HBV, HCV, or HIV positive subjects;
10. Male and female subjects of reproductive age cannot take effective contraceptive measures;
11. Pregnant or lactating women;
12. Patients with a history of mental illness or related conditions;
13. Other subjects considered unsuitable by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tissue distribution of 89Zr-NY009 | 7 days
  Biodistribution of 89Zr-NY009 evaluated by radioactive uptake values (standardized uptake values, SUVs) in various organs during repeated 89Zr-PET scans will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Chunjing Yu, Principal Investigator — Affiliated Hospital of Jiangnan University
Locations (1):
- Affiliated Hospital of Jiangnan University, Wuxi, China